CLINICAL TRIAL: NCT03651908
Title: Evaluation of Efficacy of Bioactive Silica Graft With Platelet Rich Fibrin Vs Bioactive Silica Graft Alone In The Treatment Of Intrabony Defects In Patients With Type II Diabetes Mellitus -A Randomized Clinical Study.
Brief Title: Comparison Between Bioactive Silica Graft Plus Platelet Rich Fibrin and Only Platelet Rich Fibrin Graft in Intrabony Defects With Diabetes
Acronym: CBBSGPPOPIDWD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre (Other)
Responsible Party: Principal Investigator, Dr. V. Sravanthi, PG Student, Panineeya Mahavidyalaya Institute of Dental Sciences & Research Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sravanthinovabone
Record Dates: First submitted 2018-08-23; First posted 2018-08-29 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Intrabony Periodontal Defect

STUDY DESIGN:
Intervention Model Description: In this study the patients are divided into two test groups-group A, group B. Each patient will be given careful instructions on proper oral hygiene measures. Under local anesthesia full-mouth supragingival and subgingival scaling and root planning procedure will be performed. After therapy, a periodontal evaluation will be done and the selected sites will be divided into group A and group B.
  The Group A subjects will be treated with conventional flap surgery using Bioactive silica graft with PRF as a graft.
  Group B will be treated with conventional flap surgery +bioactive silica graft alone in intrabony defects.
Who Masked: Participant
Masking Description: Sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Interventional The Group A subjects will be treated with conventional flap surgery.After reflection of the full thickness flap,the intrabony defects will be debrided and Bioactive silicate graft mixed with PRF will be used as graft material to fill the defects.
  Interventions: Procedure: Conventional Flap Surgery
- Interventional comparator (Active Comparator): Group B patients will also be treated by conventional flap surgery,employing a full thickness flap technique.The intrabony defects will be filled with Bioactive silicate only.
  Interventions: Procedure: Conventional Flap Surgery

INTERVENTIONS:
Procedure: Conventional Flap Surgery — After administering local anaesthetic a full thickness flap will be raised and reflected to expose the intrabony defects.The intrabony defects would then the debrided and grafts secured in position.Later the flap would be sutured back.
  After administering local anaesthetic a full thickness flap will be raised and reflected to expose the intrabony defects.The intrabony defects would then the debrided and grafts secured in position.Later the flap would be sutured back.

SUMMARY:
Various regenerative procedures used for the treatment of intabony defects.The Aim of this study is to compare the treatment outcome of bioactive silica graft with platelet rich fibrin Vs bioactive silica graft in the treatment of intrabony defects in patients with diabetes mellitus.

DETAILED DESCRIPTION:
Platelet rich fibrin has emerged as one of the promising regenerative material.It is a second generation platelet concentrate and is defined as an autologous leucocyte-and platelet-rich fibrin biomaterial.Platelet-rich fibrin membrane consists of a fibrin 3-D polymerized matrix in a specific structure ,with the incorporation of almost all the platelets and more than half of leucocytes along with growth factors.It enhance the stabilization and revascularization of the flaps and grafts.

Bioactive silica graft (Novabone dental putty )is being used for regenerative procedures is a premixed composite of bioactive calcium -phospho-silicate particulate which is composed solely of elements that exist naturally in normal bone (ca,p,na,si,o) and an absorbable binder which is a combination of polyethylene glycol and glycerine.Treatment of intrabony defects with bioactive silica graft has led to clinically and statistically significant probing depth reduction ,relative attachment level gain and radiographic osseous defect fill.

ELIGIBILITY:
Inclusion Criteria:

* Two or three walled defects With relative clinical attachment loss ≥3mm Probing depth≥5mm Patients with known diabetes(Type 2 hbA1c 6 to 7.4)

Exclusion Criteria:

* One wall defects Other systemically compromised patients Non- compliant patients Individuals allergic to medication Pregnant or lactating mothers Smokers

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-09-23 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Radiographic parameters - Change in bone level | Baseline and 9 months post surgery.
  Amount of bone fill in the intrabony defect (Change in bone level) to be measured by Cone Beam Computed Tomography (CBCT)

SECONDARY OUTCOMES:
clinical parameters - Changes in relative clinical attachment level | Baseline and 9 months post surgery
  Changes in relative clinical attachment level will be measured by UNC -15 probe in millimeters in the intrabony defect area

CONTACTS AND LOCATIONS:
Overall Officials: Veerendra nath Reddy, MDS, Study Director — Panineeya institute of dental sciences and research center
Locations (1):
- Panineya institute of dental sciences and research center, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Grover V, Kapoor A, Malhotra R, Uppal RS. Evaluation of the efficacy of a bioactive synthetic graft material in the treatment of intrabony periodontal defects. J Indian Soc Periodontol. 2013 Jan;17(1):104-10. doi: 10.4103/0972-124X.107484. PMID 23633783
- [Result] Sharma A, Pradeep AR. Treatment of 3-wall intrabony defects in patients with chronic periodontitis with autologous platelet-rich fibrin: a randomized controlled clinical trial. J Periodontol. 2011 Dec;82(12):1705-12. doi: 10.1902/jop.2011.110075. Epub 2011 Apr 5. PMID 21513477